CLINICAL TRIAL: NCT06376396
Title: Assessment of Combined Antiparasitic Drugs Praziquantel and Albendazole Versus Albendazole Alone in the Treatment of Active Parenchymal Neurocysticercosis in Tanzania and Zambia
Brief Title: Assessment of Combined Praziquantel and Albendazole vs Albendazole Alone to Treat Active Parenchymal Neurocysticercosis
Acronym: NeuroSolve
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: R-Evolution Worldwide S.r.l. Impresa Sociale (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); National Institute for Medical Research, Tanzania (Other Government); Sokoine University of Agriculture (Other); University of Zambia (Other); University Ghent (Other)
Responsible Party: Principal Investigator, Dario Scaramuzzi, Director, R-Evolution Worldwide S.r.l. Impresa Sociale
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101103306
Record Dates: First submitted 2024-02-25; First posted 2024-04-19 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Neurocysticercosis
Keywords: Neglected Tropical Disease; Epilepsy
MeSH Terms: conditions — Neurocysticercosis; Neglected Diseases; Epilepsy | interventions — Albendazole; Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albendazole and Praziquantel (Experimental): This arm includes combined albendazole with praziquantel, given to approximately 150 participants. Subjects will also receive dexamethasone as an adjunct treatment. An appropriate dose will be calculated per participant's body weight and administered to each participant daily for 10 days. Participants will be monitored for 30 minutes following oral medication, and a repeat dose will be administered if a participant vomits within this observation period. Additional doses (the whole cycle) will be supplied for participants failed to clear NCC in six months.
  Interventions: Drug: albendazole and praziquantel
- Albendazole (Active Comparator): This arm includes albendazole monotherapy, given to approximately 150 participants. Subjects will also receive dexamethasone as an adjunct treatment. An appropriate dose will be calculated per participant's body weight and administered to each participant daily for 10 days. Participants will be monitored for 30 minutes following oral medication, and a repeat dose will be administered if a participant vomits within this observation period. Additional doses (the whole cycle) will be supplied for participants failed to clear NCC in six months.
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: albendazole and praziquantel — Combination of albendazole plus praziquantel
  Other Names: Albendazole; Praziquantel
  Arms: Albendazole and Praziquantel
Drug: Albendazole — Albendazole alone
  Arms: Albendazole

SUMMARY:
The goal of this clinical trial is to compare the combination albendazole and praziquantel versus albendazole alone in patients affected by neurocysticercosis.

DETAILED DESCRIPTION:
This is a randomized, two arms, parallel-groups, open-label clinical trial to assess if the combination of antiparasitic praziquantel and albendazole is better than albendazole alone in the treatment of active parenchymal neurocysticercosis in Tanzania and Zambia.

Background and Study Rationale: between the forms of human cysticercosis caused by Taenia solium, neurocysticercosis is a major contributor to the burden of seizure disorders and epilepsy in most of the world, while it has relatively poor clinical evidence on treatment options, requiring further data, mainly from additional randomized controlled trials. In particular albendazole and praziquantel are the two parasiticides recommended for use in treating active neurocysticercosis (NCC). Specifically, albendazole is recommended for use in patients with a single cyst while both albendazole and praziquantel (combination therapy) are recommended for patients with multiple cysts. However, not all patients with single cysts respond to albendazole monotherapy. Combination therapy may be effective in patients with single cysts as it has already been shown effective for multiple cysts.

Most studies of treatment success for NCC have been conducted in Latin America and India. In India, the studies were performed primarily on singular cystic lesions. Despite Sub-Saharan Africa (SSA) being recognized as endemic for this parasite, no study evaluating the success of standard treatment in humans has been conducted in this region. Additionally, it is difficult to extrapolate information from other regions other than SSA due to possible differences in genetic, clinical, and environmental factors.

Primary Objective:

The primary objective of this study is to determine if the anthelmintics combination of praziquantel and albendazole is better than albendazole alone in the treatment of the active parenchymal neurocysticercosis based on cyst resolution.

Secondary Objectives:

1. To determine if the combination of antiparasitic praziquantel and albendazole is better than albendazole alone in the treatment of active parenchymal neurocysticercosis based on seizures reduction
2. To estimate the change in quality of life of patients with active symptomatic NCC before and after treatment with combined antiparasitic treatment and mono…
3. To assess the role of serology in diagnosis, management and follow up of participants treated for neurocysticercosis.

ELIGIBILITY:
Inclusion Criteria:

* Living in the study area for a continuous period of 3 years
* Adult aged 18 years and above
* Are willing and able to consent to this study
* Meet the definitions of active symptomatic NCC
* Have late onset of epilepsy or history of seizures, epileptic seizures
* Subjects willing to undergo diagnostic procedures
* Subjects medically stable enough for trial medication to be initiated
* Subjects willing to be hospitalized for 11-20 days to receive treatment for NCC
* Subjects willing to be followed up for one year following receipt of study medication

Exclusion Criteria:

* Women pregnant or breastfeeding
* Symptomatic NCC with cysts in extra-parenchymal location (sub-arachnoid and/or ventricles)
* Have uncontrolled hypertension and/or diabetes
* Have chronic consuming illness such as cancer or mental handicap to not allow them to follow the study instructions
* Have severe immunodeficiency eg. HIV/AIDS or Autoimmune diseases
* Already known allergies to albendazole or praziquantel
* Subject taking part in another clinical/pharmacological study in the 30 days preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cyst resolution or reduction in both study arms | 6 weeks and 6 months
  The primary objective of this study is to determine if the anthelmintic combination of praziquantel and albendazole is better than albendazole alone in the treatment of active parenchymal cysticercosis, based on cyst resolution. The cysts resolution is defined by at least 70% resolution at brain imaging (CT scan / MRI) between the baseline imagines and those at 6-week to 6-month following treatment.

SECONDARY OUTCOMES:
Seizures frequency | 6 weeks and 6 months
  Reduction of seizures frequency at 6-weeks to 6-months following treatment
Quality of Life questionnaire | 6 weeks, 6 months and 1 year
  The improvement in Quality of life (QoL) at 6-weeks, 6-months and 12-months following treatment.
Headache | 6 weeks, 6 months and 1 year
  The headache severity and frequency will be assessed by in-depth neurological examination, including patient-reported outcome measures (e.g. VAS - Visual Analog Scale), at the following defined time point: baseline, 6 weeks, 6 months and 1 year
Serological test results correlation with neuroimaging results | Baseline, 6 weeks, 6 months and 1 year
  To assess the role of serology in diagnosis, management and follow up of participants treated for neurocysticercosis, antigen and antibody detecting tests results will be done and the results will be compared with neuroimaging (CT/MRI), at baseline, 6-week, 6-month and 1 year following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kabemba E. Mwape, Prof., Principal Investigator — University of Zambia

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the de-identified data on efficacy and safety during publication of the study results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months after study completion.
Access Criteria: Open access

REFERENCES:
- [Background] Adebayo PB, Akinyemi RO, Ogun SA, Ogunniyi A. Seizure severity and health-related quality of life of adult Nigerian patients with epilepsy. Acta Neurol Scand. 2014 Feb;129(2):102-8. doi: 10.1111/ane.12146. Epub 2013 May 18. PMID 23682560
- [Background] Azimi A, Fattahi R, Asadi-Lari M. Knowledge translation status and barriers. J Med Libr Assoc. 2015 Apr;103(2):96-9. doi: 10.3163/1536-5050.103.2.008. No abstract available. PMID 25918490
- [Background] Fogang YF, Savadogo AA, Camara M, Toffa DH, Basse A, Sow AD, Ndiaye MM. Managing neurocysticercosis: challenges and solutions. Int J Gen Med. 2015 Oct 16;8:333-44. doi: 10.2147/IJGM.S73249. eCollection 2015. PMID 26527895
- [Background] Garcia HH, Nash TE, Del Brutto OH. Clinical symptoms, diagnosis, and treatment of neurocysticercosis. Lancet Neurol. 2014 Dec;13(12):1202-15. doi: 10.1016/S1474-4422(14)70094-8. Epub 2014 Nov 10. PMID 25453460
- [Background] Kinyanjui DW, Kathuku DM, Mburu JM. Quality of life among patients living with epilepsy attending the neurology clinic at Kenyatta National Hospital, Nairobi, Kenya: a comparative study. Health Qual Life Outcomes. 2013 Jun 18;11:98. doi: 10.1186/1477-7525-11-98. PMID 23777194
- [Background] Makasi CE, Kilale AM, Ngowi BJ, Lema Y, Katiti V, Mahande MJ, Msoka EF, Stelzle D, Winkler AS, Mmbaga BT. Knowledge and misconceptions about epilepsy among people with epilepsy and their caregivers attending mental health clinics: A qualitative study in Taenia solium endemic pig-keeping communities in Tanzania. Epilepsia Open. 2023 Jun;8(2):487-496. doi: 10.1002/epi4.12720. Epub 2023 Mar 20. PMID 36896648
- [Background] Nau AL, Mwape KE, Wiefek J, Schmidt K, Abatih E, Dorny P, Praet N, Chiluba C, Schmidt H, Phiri IK, Winkler AS, Gabriel S, Blocher J. Cognitive impairment and quality of life of people with epilepsy and neurocysticercosis in Zambia. Epilepsy Behav. 2018 Mar;80:354-359. doi: 10.1016/j.yebeh.2017.10.042. Epub 2017 Dec 6. PMID 29221763
- [Background] Nyangi C, Stelzle D, Mkupasi EM, Ngowi HA, Churi AJ, Schmidt V, Mahonge C, Winkler AS. Knowledge, attitudes and practices related to Taenia solium cysticercosis and taeniasis in Tanzania. BMC Infect Dis. 2022 Jun 13;22(1):534. doi: 10.1186/s12879-022-07408-0. PMID 35692033
- [Background] Owolabi LF, Adamu B, Jibo AM, Owolabi SD, Imam AI, Alhaji ID. Neurocysticercosis in people with epilepsy in Sub-Saharan Africa: A systematic review and meta-analysis of the prevalence and strength of association. Seizure. 2020 Jan 7;76:1-11. doi: 10.1016/j.seizure.2020.01.005. Online ahead of print. PMID 31935478
- [Background] Stelzle D, Makasi C, Schmidt V, Trevisan C, van Damme I, Welte TM, Ruether C, Fleury A, Dorny P, Magnussen P, Zulu G, Mwape KE, Bottieau E, Gabriel S, Ngowi BJ, Winkler AS; SOLID collaborators. Epidemiological, clinical and radiological characteristics of people with neurocysticercosis in Tanzania-A cross-sectional study. PLoS Negl Trop Dis. 2022 Nov 28;16(11):e0010911. doi: 10.1371/journal.pntd.0010911. eCollection 2022 Nov. PMID 36441777
- [Background] Torgerson PR, Devleesschauwer B, Praet N, Speybroeck N, Willingham AL, Kasuga F, Rokni MB, Zhou XN, Fevre EM, Sripa B, Gargouri N, Furst T, Budke CM, Carabin H, Kirk MD, Angulo FJ, Havelaar A, de Silva N. World Health Organization Estimates of the Global and Regional Disease Burden of 11 Foodborne Parasitic Diseases, 2010: A Data Synthesis. PLoS Med. 2015 Dec 3;12(12):e1001920. doi: 10.1371/journal.pmed.1001920. eCollection 2015 Dec. PMID 26633705
- [Background] Trevisan C, Damme IV, Ngowi B, Schmidt V, Stelzle D, Moller KS, Kabululu M, Makasi CE, Magnussen P, Bottieau E, Abatih E, Johansen MV, Ngowi H, Ndawi B, Mwape KE, Zulu G, Dorny P, Winkler AS, Gabriel S, On Behalf Of The Solid Consortium. Trial Design of a Prospective Multicenter Diagnostic Accuracy Study of a Point-of-Care Test for the Detection of Taenia solium Taeniosis and Neurocysticercosis in Hospital-Based Settings in Tanzania. Diagnostics (Basel). 2021 Aug 24;11(9):1528. doi: 10.3390/diagnostics11091528. PMID 34573870
- [Background] Braae UC, Saarnak CF, Mukaratirwa S, Devleesschauwer B, Magnussen P, Johansen MV. Taenia solium taeniosis/cysticercosis and the co-distribution with schistosomiasis in Africa. Parasit Vectors. 2015 Jun 12;8:323. doi: 10.1186/s13071-015-0938-7. PMID 26065414
- See also: WHO guidelines on management of Taenia solium neurocysticercosis — https://www.ncbi.nlm.nih.gov/books/NBK573855/